CLINICAL TRIAL: NCT04026282
Title: A Prospective, Randomized Controlled Study to Investigate the CLBRs of GnRH Antagonist Protocol Compared With the Standard GnRH Agonist Long Protocol for Controlled Ovarian Stimulation in Supposed Normal Ovarian Responders
Brief Title: To Investigate the Cumulative Live Birth Rates Using GnRH Antagonist or Agonist Protocol for COS in ART Treatment
Acronym: CLBR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Merck Serono GmbH, Germany (Industry); Fountain Medical Development Co., Ltd. (Industry); Guangzhou KingMed Center for Clinical Lab.Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Jie Qiao, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS700623_0020
Record Dates: First submitted 2019-02-21; First posted 2019-07-19 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Sterility
Keywords: assisted reproductive technology; live birth; fertilization
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: When patients enter this study, they will be randomly assigned to GnRH-ant group or GnRH-a group at ratio1:1 by the randomization schedule generated by a computer program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GnRH-ant protocol (Experimental): Recombinant FSH (Gonal-f®) will be administrated as routinely practiced by investigators. FSH doses will be adjusted according to the clinical experiences of investigators.The GnRH-ant (Cetrotide®) will be initiated in a fixed protocol on stimulation days 5 or 6 per the investigator's ART protocol.
  Interventions: Procedure: GnRH-ant protocol
- GnRH-a long protocol (Active Comparator): The GnRH-a (Diphereline® or Decapetyl®) 0.1mg will be administered for about 14 to 20 days for down-regulation. Gonal-f® will be administrated as routinely practiced by investigators. GnRH-a types, GnRH-a and FSH doses will be adjusted according to the clinical experiences of investigators in each site.
  Interventions: Procedure: GnRH-a long protocol

INTERVENTIONS:
Procedure: GnRH-ant protocol — Recombinant FSH (Gonal-f®) will be administrated as routinely practiced by investigators. FSH doses will be adjusted according to the clinical experiences of investigators.The GnRH-ant (Cetrotide®) will be initiated in a fixed protocol on stimulation days 5 or 6 per the investigator's ART protocol.
  Arms: GnRH-ant protocol
Procedure: GnRH-a long protocol — The GnRH-a (Diphereline® or Decapetyl®) 0.1mg will be administered for about14 to 20 days for down-regulation. Gonal-f® will be administrated as routinely practiced by investigators. GnRH-a types, GnRH-a and FSH doses will be adjusted according to the clinical experiences of investigators in each site.
  Arms: GnRH-a long protocol

SUMMARY:
This is a Phase IV, prospective, randomized controlled study to investigate the cumulative live birth rates (CLBRs) of gonadotrophin-releasing hormone (GnRH) antagonist protocol (GnRH-ant group) compared with the standard GnRH agonist long protocol (GnRH-a group) for controlled ovarian stimulation in supposed normal ovarian responders.

DETAILED DESCRIPTION:
This is a Phase IV, prospective, randomized controlled study to investigate the cumulative live birth rates (CLBRs) of gonadotrophin-releasing hormone (GnRH) antagonist protocol (GnRH-ant group) compared with the standard GnRH agonist long protocol (GnRH-a group) for controlled ovarian stimulation in supposed normal ovarian responders.

In this study, patients who are planning to undergo IVF/ICSI cycle aged ≤38 years old with normal ovarian reserve will be considered for enrollment. Approximately 888 patients will be enrolled at approximately 5 centers in China over a period of 10 months.

About 12-20 visits will be performed in this study for each patient. The CLBR with first live birth resulting from one initiated COS cycle will be compared between GnRH-a group and GnRH-ant group.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women planning to undergo IVF/ICSI cycle using conventional GnRH agonist long protocol or GnRH antagonist protocol
* Age ≤ 38 years old
* Basal AFC 8~20
* Basal FSH≤10 IU/L
* Basal E 2 <200pmol/L
* Normal uterus and at least one side of the normal ovary
* Informed consent form signed
* Willing to follow the study protocol, and able to complete this study

Exclusion Criteria:

* Previous IVF/ICSI cycles >2
* Severe hydro-salpinx (Ultrasound shows hydro salpinx﹥2cm)
* Severe endometriosis (Grade III - IV)
* Polycystic ovarian syndrome (PCOS)
* History of recurrent miscarriages (>2 times of miscarriages)
* Plan to undergo ovarian stimulation for preimplantation genetic diagnosis or preimplantation genetic screening, oocyte donation, and social or medical freezing of oocytes
* Any major systemic disease that as per Investigator's discretion precludes subject for participation in the study
* With pregnancy contraindications
* Alcoholism, drug abuse, drug addiction or patients with uncured sexually transmitted disease
* According to the judgment of the Investigator, any medical condition or any concomitant surgery/medications that would interfere with evaluation of study medications
* Simultaneous participation in another clinical study
* Plan to use urinary gonadotrophin during COS treatment

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Infertile women planning to undergo IVF/ICSI cycle aged ≤38 years old with normal ovarian reserve
Enrollment: 888 (Estimated)
Dates: Start 2018-12-27 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
the cumulative live birth rates | two years
  To investigate the cumulative live birth rates in infertile women ≤ 38 years old with normal ovarian from one initiated COS cycle.
  reserve using GnRH antagonist or agonist protocol for COS in ART treatment Numerator is the No. of women got their first live birth, the Denominator is the No. of women who attempt the ovarian stimulation.
  There will be two ways to calculate the CLBR:
  * The conservative estimate of the cumulative live birth rate, which is based on the assumption that none of the women who do not return for a subsequent embryo transfer would have had a live birth.
  * The optimal estimate of the cumulative live birth rate, which is based on the assumption that women who do not return for a subsequent embryo transfer would have had the same live birth rates as those who do return.

SECONDARY OUTCOMES:
Number of oocytes retrieved | 24 hours after Oocytes pick up
  recorded Number of oocytes retrieved on DOPU
Good-quality embryo rate (The Istanbul Consensus29) | 24 hours after Oocytes pick up
  Total the number of good quality embryos divided by Total the number of embryos
hCG positive rate | after 11 to 17 days of ET
  Numerator is the No.of β-hCG blood test which is positive results, he Denominator is the No. of β-hCG blood test. HCG test is Serum β-hCG test after 11 to 17
Implantation rate | 4 to 6 weeks after ET
  the number of gestational sacs observed divided by the number of embryos transferred
Clinical pregnancy rate | after 4 to 6 weeks of ET
  the number of clinical pregnancies expressed per 100 initiated cycles, aspiration cycles, or embryo transfer cycles. Note: When clinical pregnancy rates are given, the denominator (initiated, aspirated, or embryo transfer cycles) must be specified.
Ongoing pregnancy rate | after 12 weeks of ET
  the number of . Ongoing pregnancy divided by the number of Clinical pregnancy . Ongoing pregnancy is intrauterine pregnancy continued for 12 gestational weeks (detection of presence of gestational sac with fetal heartbeat by transvaginal ultrasound examination in week 12).
Live birth rate | two years
  Numerator is the No. of women got live birth resulting from fresh cycle (multiple births considered as one live birth), the Denominator is the No. of women who attempt the ovarian stimulation.
Cumulative clinical pregnancy rate | two years
  Numerator is the No. of women got their first clinical pregnancy, the Denominator is the No. of women who attempt the ovarian stimulation.
Miscarriage rate | after 12 weeks of ET
  the number of Miscarriage which is the natural death of an embryo or fetus before it is able to survive independently divided by the number of Clinical pregnancy .
Ectopic pregnancy rate | after 4 to 6 weeks of ET
  the number of .extrauterine pregnancy divided by the number of Clinical pregnancy .
Cycle cancelled rate and reason | On ART cycle
  Cancelled cycle is an ART cycle in which ovarian stimulation or monitoring has been carried out with the intention to treat, but which did not proceed to follicular aspiration or, in the case of a thawed embryo, to embryo transfer. Cycle cancelled rate is the number of Cancelled cycle divided by the number of embryos transferred.
severity of OHSS | two weeks after Oocytes pick up
  Assessed the severity of OHSS.
Rate of OHSS | two weeks after Oocytes pick up
  the number of OHSS divided by the number of ovum pick up. Assessed the severity of OHSS.
Time to pregnancy | 4 to 6 weeks after ET
  time from Gn Initiation to the first clinical pregnancy.
Time to live birth | nine months after pregnancy
  time from Gn Initiation to the first live birth
the Safety | Two years after signature of informed consent
  Data on AEs will be collected at scheduled and unscheduled visits, based on information spontaneously provided by the subject and/or through questioning of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Qiao Jie, Principal Investigator — Peking University Third Hospital
Locations (4):
- China (4):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The second hospital of Hebei Medical University, Baoding, Hebei
  - The third hospital of Zhengzhoui Medical University, Zhengzhou, Henan
  - Jiangsu Provincial Hospital, Nanjing, Zhejiang

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT04026282/Prot_SAP_000.pdf